CLINICAL TRIAL: NCT03739021
Title: Analgesic Requirements for Post-operative Pain Control in Total Shoulder Replacement Patients: Comparison of Interscalene Single Shot Exparel (Bupivacaine Liposome) Injections to Cervical Paravertebral Catheter With Ropivacaine (0.2% Continuous Infusion)
Brief Title: Exparel for Total Shoulder Pain
Acronym: ETSP
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37089
Record Dates: First submitted 2018-09-13; First posted 2018-11-13 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-05

CONDITIONS: Chronic Shoulder Pain
Keywords: replacement; shoulder
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: This is a randomized, open label study. A series of 60 sealed envelopes: 30 "Exparel single shot" and 30 "Ropivacaine catheter" will be blindly open for each of the 60 patients when collecting informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (30 participants) (Experimental)
  Interventions: Drug: Exparel
- Group 2 (30 participants) (Experimental)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Exparel — Single shot of the Bupivacaine Liposome, and then we follow up with patient in the recovery room with traditional common pain management. MME (milligram morphine equivalent) will be collected.
  Arms: Group 1 (30 participants)
Drug: Ropivacaine — Continuous infusion of Ropivacaine via catheter, and then we follow up with patient in the recovery room with traditional common pain management. MME (milligram morphine equivalent) will be collected.
  Arms: Group 2 (30 participants)

SUMMARY:
Total shoulder surgery (arthroplasty) is a widely successful method of treating shoulder arthritis. Although the goal of the procedure is pain relief, post-operative pain is unavoidable. Pain is a common side effect that many patients undergo while in the clinical setting and is a vital factor in influencing the length of hospital stay, narcotic usage, as well as overall patient satisfaction. Post-operative pain management typically involves elevated usage of narcotics, which is a concern among clinicians and researchers alike. To combat this issue, research is examining intraoperative procedures as a means of reducing post-operative pain scores.

Research has discovered the advantages of utilizing local anesthetic techniques as opposed to just general anesthesia. Local anesthetic blocks function by preventing the generation of nerve impulses by increasing the action-potential threshold, thereby inhibiting movement. Previous studies have demonstrated the success of local anesthetic interscalene blocks across several medical procedures. For instance, Exparel (liposomal bupivacaine) has been effective in reducing post-operative pain scores in tonsillectomy and shoulder arthroplasty. Another local anesthetic, Ropivacaine, has been found to be potent when utilized via a cervical paravertebral catheter among thoracic procedures.

Our study will compare Exparel (bupivacaine liposome) with Ropivacaine continuous infusion for post-operative pain scores in total shoulder surgery patients. Additionally, we will collect data on complications, length of stay, and other variables.

DETAILED DESCRIPTION:
Procedure Description:

The investigators commonly use these blocks for patients requiring total shoulder replacement: the patient is usually sedated with propofol. The patient is positioned in the lateral decubitus, or sitting position for this block. After the skin preparation and draping, the fingers of the non-operative hand separate the trapezius and levator scapulae muscle and a 25 gauge needle is used to anesthetize the skin and subcutaneous tissue.

The Trapezius and Levator Scapulae muscles are again separated with the non-operative hand and a 17 or 18 gauge insulated tuohy needle is inserted, which is attached to a nerve stimulator set at a current output of one to three milliamps, a frequency of two Hertz, and a pulse width of 200 to 300 microseconds. The needle is advanced towards the suprasternal notch until contact with the bony structures is made.

After contact with the bone the stylet of the needle is removed, the needle tip is walked off the bony structures in a lateral and slightly superior direction remaining on the plane of the line drawn from the dorsal spine of C6 to the suprasternal notch. After walking off of these bones structures the needle is advanced carefully in an anterior direction. As the needle is advanced there will be a motor response from the stimulator current. The muscles involved are usually the triceps, biceps, deltoids or major pectoral muscle but any muscle group of the upper limb would be acceptable for this block since the needle is now in contact with the posterior aspects of the roots of the brachial plexus. The tip of the needle at this point is situated between the anterior and middle scalene muscles and is in contact with the C6 root of the brachial plexus. At this point either a single-shot injection of Exparel will be performed, or a catheter for Ropivacaine will be inserted, as described below.

For catheter insertion: the nerve stimulator is removed from the needle and attached to the proximal end of the stimulating catheter and the tip of the catheter is inserted into the needle shaft. The nerve stimulator is usually set at a current output of one milliamp. The motor response should be unchanged. The catheter is advanced beyond the needle tip, if the motor response disappears, the catheter is careful drawn into the needle shaft and small adjustment to the needle, advancing slightly or withdrawing it slightly is done. This maneuver is repeated until the muscle twitch is unchanged during catheter advance. This indicates the catheter tip is now situated on the nerve root; the catheter is advanced 3 to 5 centimeter beyond the needle tip but not further than 5 centimeters. The needle is then removed without disturbing the catheter and the inner stylet of the catheter is also removed. The catheter position can be confirmed by attaching the nerve stimulator to the catheter, the motor response should be unchanged. The catheter is then subcutaneously tunneled and continuous infusion of Ropivacaine is inserted.

Intraoperative Management:

The intraoperative course will follow the standard of care practices. Doses/concentration of medications/agents used for the anesthetic management of the subjects enrolled in this trial may be adjusted when necessary to provide optimal subject care. Anesthesia will be induced with propofol, intravenous opioids, and other medication(s)/agent(s) at a concentration range/dose(s) based on the clinical need of the subject. Patient will be given succinylcholine to aid in intubation.

Anesthesia will be maintained in both groups with intravenous opioids, propofol and /or medication(s)/agent(s), including inhalation anesthetic agents, at a concentration range/dose(s) based on the clinical need of the subject.

Tracheal extubation will be performed at the end of anesthesia at which point the patient will be discharged to the post-anesthesia care unit.

Postoperative Management:

Upon arrival in the PACU, the (sub)investigator, using the visual analog scale, will clinically assess post-operative pain.

Assessment of patient pain levels involve a series of VAS testing postoperatively (upon arrival and every 30 minutes postoperatively until discharge from the PACU) using a 10 cm line. Patients that complain of pain intensity >5 cm/10 cm, will be given a standardized rescue intravenous dilaudid regimen, IV dilaudid at 0.4mg up to a max dose of 2mg prn q 2 hours or until a VAS of <5 is obtained. If a VAS score of <5 cannot be obtained, the PI may withdraw the patient from the study and administer another pain medication. Post-operative PACU narcotic consumption will be recorded and quantified.

All patients will be monitored with continuous pulse-oximetry. All post-operative complications will be captured.

Follow-up Period: All patients will have a planned hospital admission from the PACU. Pain will be assessed every 2 hours for the first 24 hours followed by every 4 hours until hospital discharge using the VAS scale. All post-operative complications will be captured. Post-PACU narcotic consumption will be recorded and quantified for the first 72 hours after PACU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Patients admitted to TGH for total shoulder replacement surgery
* Subjects who have given written informed consent

Exclusion Criteria:

* Patients with allergic reactions to Exparel or Ropivacaine
* Female patients who are pregnant
* Subjects known or suspected to have neuromuscular disorders impairing neuromuscular blockade (e.g., subjects with myasthenia gravis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-11-15 (Estimated)

PRIMARY OUTCOMES:
Duration of Surgery (in minutes) | Intraoperative
Post-Operative VAS Scores (10 cm scale) | 1 hour after surgery
Intraoperative Narcotics Usage (in Milligrams Morphine Equivalent; MME) | Intraoperative
Length of Post-Anesthesia Care Unit (PACU) stay (in minutes) | through study completion, 8 months-1 year (on average)
Post-Operative Narcotics Usage during PACU Stay (in Milligrams Morphine Equivalent; MME) | through study completion, 8 months-1 year (on average)
Post-Operative Narcotics Usage during first 72 hours after PACU discharge (Milligrams in Morphine Equivalents | First 72 hours after PACU discharge
Length of Hospital Stay (in hours) | through study completion, 8 months-1 year (on average)

SECONDARY OUTCOMES:
Time spent Nerve Block Procedure (in minutes) | Intraoperative
Cost of Adjuvant Therapy (in United States Dollar) | through study completion, 8 months-1 year (on average)

IPD SHARING:
Plan to Share IPD: Yes
The original records will be kept confidential. However, we will share the results of our study after removing individual identifiers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months (anticipated).
Access Criteria: upon email request

REFERENCES:
- [Background] Olson MD, Moore EJ, Price DL. A Randomized Single-Blinded Trial of Posttonsillectomy Liposomal Bupivacaine among Adult Patients. Otolaryngol Head Neck Surg. 2018 Nov;159(5):835-842. doi: 10.1177/0194599818791773. Epub 2018 Jul 31. PMID 30060719